CLINICAL TRIAL: NCT02960555
Title: Phase II Trial of Isatuximab (SAR650984) With or Without Lenalidomide in Patients With High Risk Smoldering Multiple Myeloma (ISAMAR)
Brief Title: Isatuximab With or Without Lenalidomide in Patients With High Risk Smoldering Multiple Myeloma (ISAMAR)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0148; NCI-2016-01922 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0148 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-11-08; First posted 2016-11-09 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (isatuximab) (Experimental): Patients receive isatuximab IV over 5 hours on day 1 of cycle 1, and over 3 hours thereafter on days 8, 15, and 22 of cycle 1, on days 1 and 15 of cycles 2-6, and on day 1 of subsequent cycles. Treatment repeats every 28 days for up to 30 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Isatuximab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Isatuximab — Given IV
  Other Names: Hu 38SB19; Isatuximab-irfc; SAR 650984; SAR650984; Sarclisa
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This is a multi-center, open label, phase II study designed to evaluate the efficacy of isatuximab with or without lenalidomide when given to patients with high risk smoldering multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

- To determine the rate of response according to the International Myeloma Working Group Criteria.

SECONDARY OBJECTIVES:

* To determine progression free survival (PFS) at 2 years.
* To determine overall survival (OS).
* To determine duration of response (DOR).
* To determine the clinical benefit rate (CBR).
* To evaluate safety of single agent treatment in this population
* To evaluate safety of single agent treatment in this population.
* To evaluate the immunogenicity of isatuximab.

OUTLINE:

Patients on single agent cohort receive isatuximab intravenously (IV) over 5 hours on day 1 of cycle 1, and over 3 hours thereafter on days 8, 15, and 22 of cycle 1, on days 1 and 15 of cycles 2-6, and on day 1 of subsequent cycles.

Patients on Combination Cohort with Lenalidomide receive isatuximab as in single agent cohort plus Lenalidomide po 21/28 days during cycles 1-6 only. Treatment repeats every 28 days for up to 30 cycles in the absence of disease progression or unacceptable toxicity.

Treatment repeats every 28 days for up to 30 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

-Risk factors for progression to multiple myeloma in patients with smoldering multiple myeloma (SMM) have been identified and include: percentage of bone marrow involvement by plasma cells, monoclonal spike in blood, serum free light chains in blood, presence or absence of immunoparesis in blood, percentage of normal versus abnormal plasma cells in the bone marrow compartment by using standard flow cytometry techniques and gene expression profiling of plasma cells obtained from a bone marrow aspirate.

Patients must have histologically confirmed SMM based on the following criteria. Both criteria must be met:

1. Serum monoclonal protein (IgG or IgA) ≥ 3 g/dL or urinary monoclonal protein ≥ 500 mg per 24 hours and/or clonal bone marrow plasma cells 10-60%
2. Absence of myeloma defining events or amyloidosis

Additionally, patients must meet criteria for high risk of progression to multiple myeloma by PETHEMA criteria (patients must have at least 2 risk factors present) (11):

* ≥95% abnormal plasma cells/total plasma cells in bone marrow compartment. (This is measured as a percentage of the total abnormal versus normal plasma cells in the bone marrow compartment using standard flow cytometry of the bone marrow aspirate. Having ≥95% abnormal plasma cells/total plasma cells constitutes a risk factor for progression to multiple myeloma by PETHEMA criteria)
* Immunoparesis (This term refers to the patient having low uninvolved immunoglobulins in peripheral blood, for example if a patient has IgA smoldering multiple myeloma, then either having a low IgM and/or low IgG will qualify as a risk factor for progression to multiple myeloma)

  *2 of 2 risk factors: high risk for progression at a rate of 72% at 5 years
* Creatinine clearance (CrCl) ≥ 40 ml/min. CrCl will be calculated using the Modification of Diet in Renal Disease (MDRD) equation.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of isatuximab in patients <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1.0 x 109 /L, hemoglobin more or equal than 2 grams below the institutional level of normal and platelet count ≥ 90 x 109/L. Platelet and blood transfusions are allowed on protocol. Growth factors, including granulocyte colony stimulating factors and erythropoietin are allowed.
* Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST and ALT < 3.0 x ULN.
* Females of childbearing potential and male subjects with female partners of childbearing potential must agree to avoid pregnancy by using an adequate method of contraception (2 barrier method or 1 barrier method with a spermicide or intrauterine device for 10-14 days prior to screening, during and 5 months after the last dose of isatuximab. Adequate methods of contraception are provided as examples. Other acceptable and effective methods of birth control are also permitted (eg, abstinence).
* Men must agree to not donate sperm while on the study and for at least 5 months after the last dose of isatuximab. Women of child bearing potential must have a negative serum/urine pregnancy test result within 10-14 days prior to the first administration of isatuximab and at the end of treatment visit. A negative urine pregnancy test is required prior to each subsequent isatuximab dose administration.
* Subjects must be able to give informed consent.

Exclusion Criteria:

* Evidence of myeloma defining events or biomarkers of malignancy due to underlying plasma cell proliferative disorder meeting at least one of the following(14)

  1. Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  2. Renal Insufficiency: creatinine clearance < 50 ml/min or serum creatinine > 2 mg/dL
  3. Anemia: hemoglobin value <10 g/dL or 2 g/dL < normal reference
  4. Bone lesions: one or more osteolytic lesions on skeletal radiography, computerized tomography (CT) or 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography CT (PET-CT).
  5. Clonal bone marrow plasma cell percentage ≥ 60%
  6. Involved: uninvolved serum free light chain ratio ≥100 measured by Freelite assay (The Binding Site Group, Birmingham, UK)
  7. >1 focal lesions on MRI studies (each focal lesion must be 5 mm or more in size)
* Bisphosphonates are permitted, including pamidronate, zoledronic acid, alendronate, ibandronate, risedronate.
* Treatment with corticosteroids is not permitted, unless the patient is on a stable chronic dose of inhaled steroids to treat respiratory diseases or on stable chronic steroid replacement therapy for endocrinology disorders.
* Radiotherapy is not permitted.
* Prior or concurrent treatment for smoldering multiple myeloma with chemotherapy agents approved for the treatment of smoldering multiple myeloma or CD38 drugs is not permitted.
* Plasma cell leukemia
* Pregnant or lactating females. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with isatuximab, breastfeeding should be discontinued if the mother is treated with isatuximab. These potential risks may also apply to other agents used in this study.
* Active hepatitis B or C infection
* Known HIV infection
* Intolerance to infused protein products, sucrose, histidine or polysorbate 80
* Concurrent treatment with other anti-cancer therapy is not permitted
* Patients must not have uncontrolled intercurrent illness including hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia. Patients should not have New York Heart Association classification III or IV heart failure at baseline.
* Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance with study requirements
* Contraindication to any concomitant medication, including pre-medications or hydration given prior to therapy
* Major surgery within 1 month prior to enrollment
* Patients with pre-existing pulmonary uncontrolled disease will be excluded. Uncontrolled refers to patients having had at least one hospitalization due to pulmonary disease (for example, asthma, chronic obstructive pulmonary disease) within the 6 months prior to enrollment in the study. Patients with previous history of pneumonitis will be excluded.
* Recruitment Strategies
* Patients that are seen in clinic at MD Anderson, Memorial Sloan Kettering Cancer Center and Mount Sinai meeting eligibility criteria will be screened for the protocol
* Other participant sources will be from outside physician referrals.
* Our outside physician referral network has a high representation of minorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall response (>= partial response) | 6 months
  The trial will be conducted by the Simon's optimal two-stage design and the response rate will be estimated accordingly. Summary statistics will be provided for continuous variables. Frequency tables will be used to summarize categorical variables. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate and the adverse event rate.

SECONDARY OUTCOMES:
Progression free survival | 2 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Overall survival | Up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Incidence of adverse events | Up to 5 years
  Adverse events will be summarized by frequency tables for all patients. For the safety endpoint, per-treated analysis will be performed to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.

OTHER OUTCOMES:
Rate of minimal residual disease (MRD) negativity at complete remission assessed by flow cytometry and next generation sequencing | Up to 2 years
  MRD assessed will be based on bone marrow aspirates. Will use 8-color flow cytometry as well as next generation sequencing of the variable (V) diversity (D) joining (J) segment.
Molecular profiling | Baseline up to progression of disease, assessed up to 5 years
  Will include whole exome sequencing and gene expression profiling and cellular (including flow cytometry) profiling using bone marrow aspirate samples.
Immune characterization | Baseline up to 2 years
  Cell surface and functional studies of dendritic, T-, B-, natural killer (NK)- and NKT-cells using bone marrow aspirate samples and peripheral blood samples.
Mechanisms of resistance to isatuximab | Up to 5 years
  Will include generation of isatuximab resistant myeloma cells, gene expression profiling in drug-naive and resistant myeloma cells, identification of molecular pathways involved in the generation of the resistant phenotype and mechanisms of dual resistance to isatuximab and other myeloma drugs.
Genetic polymorphisms | Baseline
  Will include FcGR genetic variations assessed using peripheral blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Sheeba Thomas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org